CLINICAL TRIAL: NCT06710483
Title: Do Telehealth Dental Interviews Facilitate in Person Clinical Visits for Patients With Complex Medical Needs?
Brief Title: A Pilot Project to Facilitate Dental Care and Reduce Barriers For Youth With Disabilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Deborah Munroe Noonan Memorial Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-45236; 55211805 (Other Grant/Funding Number: Deborah Munroe Noonan Memorial Research Fund)
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Intellectual Disability, Variable
Keywords: Intellectual and developmental disabilities; Telehealth interview; Pediatric dental care; Pre-Dental Care Telehealth Visit
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Dental Visit Telehealth Interview (Experimental): Participants randomized into this arm will receive a scripted telehealth interview before the scheduled dental visit.The participant's' caregiver and dentist will complete a survey within a week of the dental visit.
  Interventions: Behavioral: Pre-Dental Telehealth (PDT)
- Routine Dental Visit (No Intervention): Participants randomized into this arm will receive standard of care dental visit. The participant's' caregiver and dentist will complete a survey within a week of the dental visit.

INTERVENTIONS:
Behavioral: Pre-Dental Telehealth (PDT) — The PDT will be a scripted telehealth interview 3-7 days before the scheduled dental visit to review medical and dental history, to evaluate the participants' needs for the dental visit, and to set an agreed goal for the dental visit using shared decision making. The goal wlll be one of the following: Goal 1: exam cleaning only, Goal 2: exam and cleaning, Goal 3: exam, radiographs, and cleaning.
  Arms: Pre-Dental Visit Telehealth Interview

SUMMARY:
This randomized clinical trial is an innovative pilot project to determine the acceptance and impact of telehealth visits on youth with intellectual and developmental disabilities (IDD), their caregivers, and dentists. The impact of the telehealth visit will be assessed by: 1) determining if the intervention group was more likely to achieve the set goals and 2) Likert scaled surveys of satisfaction of caregivers and dentists. Qualitative data will be collected to inform improvement on clinical interviews by the dentist.

ELIGIBILITY:
Inclusion Criteria:

* Have an appointment for a routine check up at the Pediatric Clinic or Pediatric Health Center at the Boston University Goldman School of Dental Medicine
* Diagnosis of Intellectual or developmental disability (IDD)
* Have a caregiver who is willing to participate in the study
* Have a dental provider who is willing to participate in the study
* English speaking

Exclusion Criteria:

* None

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants who successfully completed the dental visit goal | within 1 week of the dental visit
  This will be assessed by reviewing the goal set in the PDT and comparing it to what was done at the dental visit.

SECONDARY OUTCOMES:
Caregiver satisfaction | within 1 week of the dental visit
  This outcome will be assessed by analyzing the 10 Likert scale items from a 13-item investigator developed survey. Each off the 10 items is answered with a 5 response Likert scale [Strongly disagree, Disagree, Neither Disagree nor Agree, Agree, Strongly Agree].
Dentist satisfaction | within 1 week of the dental visit
  This outcome will be assessed by analyzing the 10 Likert scale items from a 12-item investigator developed survey. Each off the 10 items is answered with a 5 response Likert scale [Strongly disagree, Disagree, Neither Disagree nor Agree, Agree, Strongly Agree].

CONTACTS AND LOCATIONS:
Overall Officials: Keri Discepolo, DDS MPH, Principal Investigator — Goldman School of Dental Medicine
Locations (1):
- Goldman School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No